CLINICAL TRIAL: NCT01658462
Title: A Phase II Randomized Study of Docetaxel With or Without NINTEDANIB (BIBF-1120) in Patient Receiving a First or Second-line of Chemotherapy for HER Negative Metastatic or Locally Recurrent Breast Cancer
Brief Title: Phase II Study of Docetaxel +/- Nintedanib in Breast Cancer
Acronym: VAROCE-1206
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAROCE - 1206; 2012-002214-38 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-07 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: locally recurrent or metastatic breast cancer; Docetaxel; Nintedanib
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Docetaxel + Nintedanib
  Interventions: Drug: Docetaxel; Drug: Nintedanib
- Arm B (Active Comparator): Docetaxel + increase of the dose
  Interventions: Drug: Docetaxel; Drug: Docetaxel: increase of the dose

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 IV Day 1 / 3 weeks
  Other Names: Taxotere
Drug: Nintedanib — 200 mg x 2 per os daily from D2*
  *No Nintedanib on days when docetaxel is administered
  Other Names: OFEV
  Arms: Arm A
Drug: Docetaxel: increase of the dose — Dose can be increased to 100 mg/m² secondarily at cycle 2 on the initiative of the investigator
  Other Names: Taxotere
  Arms: Arm B

SUMMARY:
National, randomized, unblinded, phase IIb trial with 2 strata: First-line chemotherapy / Second-line chemotherapy for locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
Patients will be stratified at randomization according to first-line chemotherapy / Second-line chemotherapy for metastatic or locally recurrent breast cancer

Treatment until progression or unacceptable toxicity Visits are planned every 3 weeks during treatment and every 3 months after end of treatment or patient's withdrawal

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Histologically or cytologically confirmed adenocarcinoma of the breast
* Locally recurrent or metastatic disease
* HER 2 negative status
* Requiring a first or a second-line chemotherapy for locally recurrent or metastatic disease.
* Prior first line chemotherapy not containing Docetaxel
* Measurable or evaluable disease according to RECIST 1.1 criteria
* Allowed prior chemotherapy as follows :

  * Docetaxel in the neoadjuvant or adjuvant setting is allowed provided that relapse has been observed more than 12 months after the end of docetaxel treatment
  * Bevacizumab in 1st line is allowed with a wash-out of 4 weeks, with recovery to NCI-CTCAE v3.0 toxicity
* ECOG performance status 0-1
* Adequate bone marrow, hepatic and renal functions as evidence by the following:

  * Hemoglobin ≥ 10 G/100 mL
  * Neutrophils count ≥ 1500 /mm3
  * Platelets ≥ 100 000 /mm3
  * Total bilirubin ≤ ULN (ULN:Upper Limit of Normal)
  * SGOT/SGPT ≤ 1.5 x ULN (≤ 2.5 x ULN in case of hepatic metastasis)
  * Serum alkaline phosphatase ≤ 2.5 x ULN
  * Creatinin clearance ≥ 45 ml/min or creatinin ≤ 1.5 x ULN
  * Proteinuria < CTCAE grade 2
* Coagulation parameters: International normalised ratio (INR) ≤ 2, prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 50% of deviation of institutional ULN
* Effective contraception for patients (male and female) with reproductive potential during their entire participation in the study and during 3 months after the last administration of Nintedanib or Docetaxel
* Negative pregnancy test (serum beta-HCG) performed within 1 week prior to start of study treatment in females with reproductive potential
* Patient covered by government health insurance
* Signed and dated written informed consent prior to admission to the study in accordance with ICH-GCP guidelines and to the local legislation

Exclusion Criteria:

* Concomitant hormone therapy for metastatic breast cancer
* Patients with dysphagia, or inability to swallow the tablets
* Other serious illness or medical conditions: Cardiac disease
* Unstable diabetes
* Uncontrolled hypercalcemia
* Pregnancy or breast feeding woman
* Unable for medical follow-up (geographic, social or mental reasons)
* Prior treatment with Nintedanib or any other VEGFR inhibitor
* Known hypersensitivity to the trial drugs , to their excipients, to peanut, to soya or to contrast media
* Contra indication to the use of the backbone treatment and to the comparator
* Active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before randomisation)
* Leptomeningeal disease
* Radiographic evidence of cavitary or necrotic tumors
* Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels
* History of clinically significant haemorrhagic or thromboembolic event in the past 6 months
* Known inherited predisposition to bleeding or thrombosis
* Significant cardiovascular diseases ( i.e. uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > NYHA II, serious cardiac arrhythmia, pericardial effusion)
* Other malignancies within the past 5 years other than basal cell skin cancer or carcinoma in situ of the cervix
* Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy
* Active or chronic hepatitis C and/or B infection
* Active alcohol or drug abuse
* Significant weight loss (> 10% of BW) within past 6 months prior to inclusion into the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12-31 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) in patients receiving Docetaxel + Nintedanib treatment (Arm A) compared to Docetaxel alone (Arm B) | baseline, every 9 weeks (or 3 cycles), up to 6 months
  6-months progression free disease

SECONDARY OUTCOMES:
response rate | baseline, every 9 weeks (or 3 cycles), up to 6 months
  according to RECIST 1.1
overall survival | up to 2 years
  time from the date of randomization to the date of death from any cause
quality of life by QLQ-C30 and additionnel module BR23 | baseline, every 9 weeks (or 3 cycles), up to 6 months
  questionnaire : EORTC QLQ C30 (Additional module BR23)
biological markers levels in tumors and endothelial cells | baseline, every 9 weeks (or 3 cycles), up to 6 months
  biological analysis of cells RT-qPCR analysis, including endothelial cells using a specific reference gene
biological markers in patient serum | baseline, every 9 weeks (or 3 cycles), up to 6 months
  biological analysis in patient's serum Dosage of VEGF-A, -C, FGF-1, -2, PDGF-AA, -AB, -BB in patient's serum
safety profile of Nintedanib | before each cycle, 3 weeks after the last dose or at the end of study
  according to NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jacques BONNETERRE, MD PhD, Study Director — Oscar Lambret Center
Locations (12):
- France (12):
  - CHU Amiens- Hôpital Sud, Amiens
  - Hôpital Privé les Bonnettes, Arras
  - Centre Pierre Curie, Beuvry
  - CH Compiègne-Noyon, Compiègne
  - Centre Léonard de Vinci, Dechy
  - Centre Oscar Lambret, Lille
  - Polyclinique de Limoges - site Chénieux, Limoges
  - Institut Jean Godinot, Reims
  - CMCO de la Côte d'Opale, Saint-Martin-Boulogne
  - Hôpital Bretonneau, Tours
  - Nouvelle Clinique des Dentellières, Valenciennes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No